CLINICAL TRIAL: NCT01964092
Title: Effect Evaluation of Individual Placement and Support (IPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IPS-NAV
Record Dates: First submitted 2013-07-17; First posted 2013-10-17 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Psychosis; Substance Abuse; Depression; Anxiety
Keywords: Disability; Individual placement and support; Mental health; Quality of life; Randomized controlled trial; Rehabilitation; Return to work; Supported employment
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Depression; Anxiety Disorders; Psychological Well-Being | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Placement and Support (Experimental): Individual Placement and Support (IPS) is a well-defined intervention aiming to help people with disabilities participate in the competitive labor market by working in jobs they prefer with the professional help that they need. IPS actively facilitates job acquisition and provides ongoing support once the client is employed.
  Interventions: Behavioral: Individual Placement and Support
- Ordinary employment schemes (Active Comparator): The control group will receive treatment as usual in terms of the ordinary employment schemes offered to this group, primarily Work with assistance and/or Traineeship in a sheltered business.
  Interventions: Behavioral: Ordinary employment schemes

INTERVENTIONS:
Behavioral: Individual Placement and Support
  Arms: Individual Placement and Support
Behavioral: Ordinary employment schemes
  Arms: Ordinary employment schemes

SUMMARY:
Roughly one third of disability pensions issued in Norway are classified as mental and behavioral disorders. The proposed study aims to evaluate the effect of an innovative intervention for returning people with moderate to severe mental health disorders to work: Individual Placement and Support (IPS).

DETAILED DESCRIPTION:
The current employment schemes offered to this diagnostic group are primarily based on a train-and-place principle with assisted or sheltered employment. Building on a place-and-train principle, rather, the IPS model of supported employment in real-life competitive work settings has proven largely successful in previous studies, but has never been tested in this group in the Norwegian context.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be undergoing treatment for moderate to severe mental health problems.
* Participants must have an expressed desire to work.
* Participants must have sufficient Norwegian reading and writing skills.

Exclusion Criteria:

* Participants are not undergoing treatment for moderate to severe mental health problems.
* Participants do not have an expressed desire to work.
* Participants do not have sufficient Norwegian reading and writing skills.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Reme, PhD, Study Director — NORCE Norwegian Research Centre AS
Locations (1):
- Uni Research, Bergen, Norway

REFERENCES:
- [Background] Sveinsdottir V, Lovvik C, Fyhn T, Monstad K, Ludvigsen K, Overland S, Reme SE. Protocol for the effect evaluation of Individual Placement and Support (IPS): a randomized controlled multicenter trial of IPS versus treatment as usual for patients with moderate to severe mental illness in Norway. BMC Psychiatry. 2014 Nov 18;14:307. doi: 10.1186/s12888-014-0307-7. PMID 25403470
- [Derived] Fyhn T, Ludvigsen K, Reme SE, Schaafsma F. A structured mixed method process evaluation of a randomized controlled trial of Individual Placement and Support (IPS). Implement Sci Commun. 2020 Oct 30;1:95. doi: 10.1186/s43058-020-00083-9. eCollection 2020. PMID 33145494
- [Derived] Reme SE, Monstad K, Fyhn T, Sveinsdottir V, Lovvik C, Lie SA, Overland S. A randomized controlled multicenter trial of individual placement and support for patients with moderate-to-severe mental illness. Scand J Work Environ Health. 2019 Jan 1;45(1):33-41. doi: 10.5271/sjweh.3753. Epub 2018 Aug 2. PMID 30074050
- See also: Study website — http://uni.no/nb/uni-helse/stress-helse-og-rehabilitering/effektevaluering-av-individuell-jobbsttte-ips-2/

RESULTS

PARTICIPANT FLOW:
Groups:
- Individual Placement and Support: Individual Placement and Support (IPS) is a well-defined intervention aiming to help people with disabilities participate in the competitive labor market by working in jobs they prefer with the professional help that they need. IPS actively facilitates job acquisition and provides ongoing support once the client is employed.
  Individual Placement and Support
- Ordinary Employment Schemes: The control group will receive treatment as usual in terms of the ordinary employment schemes offered to this group, primarily Work with assistance and/or Traineeship in a sheltered business.
  Ordinary employment schemes
Period: Overall Study
Arm/Group | Individual Placement and Support | Ordinary Employment Schemes
Started | 229 | 181
Completed | 227 | 181
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Placement and Support | Ordinary Employment Schemes | Total
Number analyzed (Participants) | 229 | 181 | 410
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 229 | 181 | 410
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.86 (10.81) | 34.77 (10.76) | 34.82 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 85 | 199
  Male | 115 | 96 | 211
Region of Enrollment [Number; unit: participants]
  Norway | 229 | 181 | 410

OUTCOME MEASURES:

1. Primary Outcome: Labor Market Participation in Ordinary Paid Employment, or Education.
Description: Labor market participation is operationalized as being registered in the Norwegian Labour and Welfare Administrations (NAV) State Register of Employers and Employees, and not as a recipient of unemployment or sickness benefits, not receiving work assessment allowance or disability pension with a higher degree of disability than by study inclusion, and registered yearly income.
Time Frame: 1 year (2016)
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Placement and Support | Ordinary Employment Schemes
Number analyzed (Participants) | 227 | 181
Participants | 83 | 49

ADVERSE EVENTS:
Time Frame: During the follow-up period, 0-18 months.
Description: The follow-up which was offered to participants has not been led to adverse events in the current nor previous studies, as it does not pose specific threats or risks to participants.
Arm/Group | Individual Placement and Support | Ordinary Employment Schemes
All-Cause Mortality (participants affected / at risk) | 2/227 | 0/181
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/181
Other Adverse Events (participants affected / at risk) | 0/227 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No